CLINICAL TRIAL: NCT05394844
Title: Study of a Culturally Tailored Diabetes Education Curriculum With Real-time Continuous Glucose Monitoring in a Latinx Population With Type 2 Diabetes (The CUTDM With CGM Study)
Brief Title: Diabetes Education With Real-time Continuous Glucose Monitoring
Acronym: CUTDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: American Diabetes Association (Other); Washington State University (Other); Sea Mar Community Health Centers (Other); DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, Nicole Ehrhardt, Assistant Professor of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00014396
Record Dates: First submitted 2022-04-19; First posted 2022-05-27 (Actual); Results first posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Type 2
Keywords: continuous glucose monitoring; diabetes education
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Real Time Continuous Glucose Monitoring using Dexcom G6 and Diabetes education
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- CGM with DM education (Active Comparator): if you are in the intervention group you will received culturally tailored diabetes education and use a Real Time CGM device to see your glucose over 12 weeks. Both group will completed blinded CGM at the beginning of the study and at 24 weeks
  Interventions: Device: Dexcom G6
- Education only (No Intervention): If you are in the control group your will receive culturally tailored diabetes education and wear a blinded prior to education and after education sessions complete and 24 weeks

INTERVENTIONS:
Device: Dexcom G6 — Dexcom G6 CGM device
  Other Names: Compañeros en Salud (Partners in Health) curriculum
  Arms: CGM with DM education

SUMMARY:
Determine the impact of the Compañeros en Salud (Partners in Health) curriculum in conjunction with RT-CGM on glycemic control in Latinx patients with T2D. Participants will be randomized to receive the Companeros en Salud diabetes self-management education and support (DSMES) intervention with or without RT-CGM

DETAILED DESCRIPTION:
The prevalence of type 2 diabetes is increasing especially in the Latinx community and in family members of those already living with diabetes. Diabetes education is a cornerstone of treatment but is often not culturally tailored and there is limited data on benefit of virtual delivery of sessions. Real Time Continuous glucose monitoring is a tool to improve diabetes but is not readily available to those living with type 2 diabetes not on multiple doses of insulin. Furthermore here is little to no data on RT-CGM use in different minority populations. Data is also lacking on if diabetes education for an individual affects the family unit. We hypothesize that culturally tailored Diabetes self-management education using and support (DSMES) using a team approach of health educators and Community health workers will improve glycemic indices. We further hypothesis that RT-CGM coupled to DSMES will enhances glycemic benefit and change nutrition and activity behaviors. This will be a randomized control trial of 100 Latinx participants who will all receive culturally tailored DSMES with or without cycle RT-CGM over 12 weeks. Primary outcome will be mean A1C improvement at 12 and 24 weeks based on attendance of sessions and RT-CGM use. Secondary outcomes will be satisfaction with education and CGM, changes in weight, blood pressure and self-reported nutrition and exercise changes. This study will be the first study to examine how DSMES with and without RT-CGM use improves health outcomes in the Latinx population and their families

ELIGIBILITY:
Inclusion Criteria:

1. Participants adults 18-60 years old
2. Self-identify as Latinx
3. Have had a clinical diagnosis of T2D within the last 15 years with or without medication use
4. Have an A1C ≥8.0% at screening
5. Own or have routine access to a personal device that allows attending educational sessions virtually
6. Be physically and cognitively able to use the home CGM monitoring device
7. Be willing and able to follow all other study procedures

Exclusion Criteria

* Exclusion Criteria.

  1. Duration of diabetes >15 years
  2. Type 1 diabetes or latent autoimmune diabetes
  3. Current use of prandial insulin
  4. Any condition that prevents walking at least 1 city block
  5. History of serious mental illness other than adequately treated depression
  6. History of bariatric surgery or current participation in a weight management program
  7. Current diagnosis of cancer or other serious or systemic medical condition
  8. Significant active cardio- or cerebrovascular disease after review by PI
  9. Pregnancy
  10. know history x of of hypoglycemia unawareness
  11. Unable to read, understand, and sign the Informed Consent Form (ICF) and if applicable, an Authorization to Use and Disclose Protected Health Information form (consistent with Health Insurance Portability and Accountability Act of 1996 [HIPAA] legislation), communicate with the investigator, and understand and comply with protocol requirements

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-11-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Washington Diabetes Institute, Seattle, Washington
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ehrhardt N, Cedeno B, Montour L, Sinclair K, Ferguson G, Berberian P, Comstock B, Wright L. Effectiveness of a culturally tailored diabetes education curriculum with real-time continuous glucose monitoring in a Latinx population with type 2 diabetes: the CUT-DM with CGM for Latinx randomised controlled trial study protocol. BMJ Open. 2023 Dec 28;13(12):e082005. doi: 10.1136/bmjopen-2023-082005. PMID 38154895

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CGM With DM Education | Education Only
Started | 61 | 59
Completed | 45 | 40
Not Completed | 16 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CGM With DM Education | Education Only | Total
Number analyzed (Participants) | 61 | 59 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (9) | 47 (7) | 46 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 24 | 53
  Male | 32 | 35 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 61 | 59 | 120
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 61 | 59 | 120
income less than 49,999 [Number; unit: participants] | 35 | 39 | 74
preferred primary language spanish [Number; unit: participants] | 59 | 58 | 117
education highschool or less [Number; unit: participants] | 55 | 54 | 109
insurance- self pay [Count of Participants; unit: Participants] | 44 | 36 | 80

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1C
Description: Percent change in A1C
Time Frame: change at 12 weeks
Population: change in A1c over 12 weeks
Measure: Mean (95% Confidence Interval); unit: percent change in A1C
Arm/Group | CGM With DM Education | Education Only
Number analyzed (Participants) | 41 | 40
percent change in A1C | -2.3 [-3.1 to -1.5] | -1.5 [-2.3 to -0.6]

2. Secondary Outcome: CGM Mean Glucose
Description: mean glucose at 12 weeks
Time Frame: 12 weeks
Population: those that had baseline and 12 week CGM data
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | CGM With DM Education | Education Only
Number analyzed (Participants) | 45 | 38
mg/dl | 208.4 (62.5) | 239.6 (84.4)

3. Secondary Outcome: CGM Percentage of Time in Range
Description: percentage of time in range( tir)
Time Frame: 12 WEEKS
Population: THOSE WITH CGM DATA AVAILABLE AT 12 WEEKS
Measure: Mean (95% Confidence Interval); unit: percentage of tir
Arm/Group | CGM With DM Education | Education Only
Number analyzed (Participants) | 45 | 38
percentage of tir | 13.2 [1.3 to 25.2] | 6.2 [-6.7 to 19.1]

4. Secondary Outcome: Percent Change in BMI
Description: percent change BMI ((kg/m2)
Time Frame: change at 12 WEEKS
Population: THOSE WITH 12 WEEKS BMI AVAILABLE
Measure: Mean (95% Confidence Interval); unit: % bmi CHANGE
Arm/Group | CGM With DM Education | Education Only
Number analyzed (Participants) | 41 | 40
% bmi CHANGE | -1 [-6.6 to 8.6] | -2.4 [-10 to 5.3]

5. Secondary Outcome: Blood Pressure Systolic
Description: change in blood pressure
Time Frame: change at 12 WEEKS
Population: those with blood pressure available 12 weeks
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | CGM With DM Education | Education Only
Number analyzed (Participants) | 41 | 40
mmHg | -2.5 [-9.3 to 4.4] | -0.3 [-7.2 to 6.7]

6. Secondary Outcome: Physical Activity Questionnaire IPAQ
Description: increase or decrease in days of vigorous activity - one question in IPAQ.
Time Frame: 12 weeks
Population: THOSE WITH questionnaire Available 12 weeks
Measure: Mean (Standard Deviation); unit: number of days
Arm/Group | CGM With DM Education | Education Only
Number analyzed (Participants) | 41 | 40
number of days | 1 (3.8) | 0.14 (1.45)

7. Secondary Outcome: International Physical Activity Prevalence Study SELF-ADMINISTERED ENVIRONMENTAL MODULE(PANES):
Description: Question Neighborhood Questionnaire/Neighborhood Safety questions 1
  1. In general, how do you feel about your neighborhood? Do you feel it's a very bad, a fairly bad, a fairly good, or a very good place to live?
  reported number that felt it was very bad or fairly bad
Time Frame: baseline
Population: those that completed survey and felt bad or fairly bad about neighborhood
Measure: Count of Participants; unit: Participants
Arm/Group | CGM With DM Education | Education Only
Number analyzed (Participants) | 61 | 58
Participants | 3 | 9

8. Secondary Outcome: PHQ9 Depression Score- Those With PHQ9>15
Description: Scores less than 5 almost always signified the absence of a depressive disorder; scores of 5 to 9 predominantly represented patients with either no depression or subthreshold (i.e., other) depression; scores of 10 to 14 represented a spectrum of patients; and scores of 15 or greater usually indicated major depression.
Time Frame: 12 weeks
Population: those that completed questionnaire are 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | CGM With DM Education | Education Only
Number analyzed (Participants) | 41 | 40
Participants | 5 | 7

9. Secondary Outcome: PAID-5 Problem Areas in Diabetes Those With Score > 8
Description: the scale gives a total score from 0 to 20. A score of 8 and above indicates a high level of diabetes-related distress
Time Frame: score at 12 weeks
Population: those with questionnaire available at 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | CGM With DM Education | Education Only
Number analyzed (Participants) | 41 | 40
Participants | 13 | 11

10. Secondary Outcome: Self-care for Diabetes (SDSCA) Number of Days Reporting Self Care
Description: The Summary of Diabetes Self-Care Activities asks patient about diabetes self-care activities during the past 7 days and for each activity they can answer 0 days out of the week to a max of 7 days out of the week with higher score indicating more days doing this self -care activity and positive results
Time Frame: composite score at 12 weeks
Population: those with questionnaire available at 12 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CGM With DM Education | Education Only
Number analyzed (Participants) | 41 | 40
days | 5.3 (2.04) | 3.3 (2.18)

11. Secondary Outcome: Modified Joslin Diabetes Center CGM Experience
Description: Experiences of CGM @Joslin 2009 scale range from 5 (strongly agree) to 1 ( strongly disagree) statements/questions that measured the amount of satisfaction that was derived from use of continuous glucose monitoring. Higher score meant perceived benefit/ better outcome
Time Frame: 12 weeks
Population: participant who completed questionnaire and wore real-time CGM
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CGM With DM Education
Number analyzed (Participants) | 41
score on a scale | 4.33 (0.55)

12. Secondary Outcome: Perception of Behavior Modification After Real-Time- CGM Use
Description: Did use of Real-Time- cgm in intervention group contribute to a healthier lifestyle ? yes
Time Frame: at 12 weeks
Population: particpants who completed questionnaire
Measure: Count of Participants; unit: Participants
Groups:
- Real Time- CGM With DM Education: if you are in the intervention group you will received culturally tailored diabetes education and use a Real Time CGM device to see your glucose over 12 weeks. Both groups will completed blinded CGM at the beginning of the study and at 24 weeks
  Dexcom G6: Dexcom G6 CGM device
Arm/Group | Real Time- CGM With DM Education
Number analyzed (Participants) | 37
Participants | 36

13. Secondary Outcome: Household/Family Member Perception of Lifestyle Changes
Description: household members perception of lifestyle changes after family member participated in education with CGM. Overall, do you feel Continuous Glucose Monitoring contributed to your making changes for a healthier lifestyle? yes
Time Frame: 12 weeks
Population: number of household members that completed the survey
Measure: Count of Participants; unit: Participants
Groups:
- CGM With DM Education Household Member: intervention group household member received culturally tailored diabetes education and used a Real Time CGM device to see your glucose over 12 weeks.
  Dexcom G6: Dexcom G6 CGM device
Arm/Group | CGM With DM Education Household Member
Number analyzed (Participants) | 15
Participants | 13

14. Secondary Outcome: Pedometer
Description: average number of steps per day
Time Frame: at 12 weeks
Population: those that had pedometry data at 12 weeks
Measure: Mean (Standard Deviation); unit: number of steps per day
Arm/Group | CGM With DM Education | Education Only
Number analyzed (Participants) | 14 | 14
number of steps per day | 6931 (3680) | 4703 (1567)

15. Secondary Outcome: Self-Efficacy for Diabetes
Description: the scale is 1-10 and the score is the mean of the eight items. If more than two items are missing, do not score the scale. Higher number indicates higher self-efficacy
Time Frame: score at 12 weeks
Population: those that completed survey at 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CGM With DM Education | Education Only
Number analyzed (Participants) | 41 | 40
units on a scale | 8.5 (1.4) | 7.7 (1.6)

16. Secondary Outcome: Food Insecurity Short Form 6 Question Composite With Score Reported as a Composite: High or Marginal Food Security, Low Food Security, Very Low Food Security
Description: number of participants that had high or marginal food security based on 6 questions (geared to assess access or lack of access to food) composite score
Time Frame: baseline
Population: those that completed survey
Measure: Count of Participants; unit: Participants
Arm/Group | CGM With DM Education | Education Only
Number analyzed (Participants) | 61 | 58
Participants | 30 | 37

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | CGM With DM Education | Education Only
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/59
Other Adverse Events (participants affected / at risk) | 0/61 | 0/59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-10): https://cdn.clinicaltrials.gov/large-docs/44/NCT05394844/Prot_SAP_004.pdf
  • Informed Consent Form (2023-02-22): https://cdn.clinicaltrials.gov/large-docs/44/NCT05394844/ICF_005.pdf